CLINICAL TRIAL: NCT06512792
Title: Mobile App-Based Remote Management Model for IBD Patients: A Multi-Center Randomized Controlled Study
Brief Title: Mobile App-Based Remote Management Model for IBD Patient
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CHEC2024-210
Record Dates: First submitted 2024-02-18; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Telemedicine; Mobile APP; Inflammatory Bowel Disease; Daily Management; Disease Activity; Randomized controlled
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: IBD patients meeting the inclusion criteria will be stratified and randomly assigned to either the intervention group or the control group. Participants in the intervention group will undergo remote healthcare management by the researchers through the WeChat platform, including the establishment of electronic health records, health management monitoring, risk warning and intervention, and health education. On the other hand, participants in the control group will receive no specific guidance and will only receive standard traditional treatment services (i.e., medication according to prescription and routine outpatient follow-ups).Colonoscopy will be required for endoscopic assessment at baseline and at the 12-month follow-up. Additionally, participants will be surveyed monthly for one year to assess the utilization of healthcare resources. At the baseline, 6-month, and 12-month visits, researchers will evaluate disease activity, quality of life , and healthcare resource utilization.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients undergoing telemedicine interventions (Experimental): Participants in the intervention group received telemedicine management from researchers through the mobile app platform (establishing electronic health records, health management monitoring, risk warning and intervention, health education).
  Interventions: Behavioral: Telemedicine management through Mobile APP
- IBD patients receiving traditional medical care (No Intervention): The control group received no guidance and only standard traditional care services (i.e., prescribed medication and regular outpatient follow-up).

INTERVENTIONS:
Behavioral: Telemedicine management through Mobile APP — According to the patient's electronic health records, each participating center researcher conducts personalized medication reminders and follow-up reminders for enrolled patients on a one-on-one basis. Simultaneously, patients are advised to monitor their health at home, regularly record and upload changes in clinical symptoms, medication, diet, exercise, etc., on the Mobile APP platform. Periodically, self-assessment scales are distributed through the Questionnaire Star platform to assess and record the patient's disease activity, quality of life, sleep, psychological status, etc., and update the information in the electronic health records.Based on the patient's clinical symptoms, self-assessment scales, and feedback from medical institution tests and examinations, each participating center researcher will promptly assess potential health risks, send warning alerts, and provide targeted informational support and interventions.
  Arms: Patients undergoing telemedicine interventions

SUMMARY:
Inflammatory Bowel Disease (IBD) is a chronic inflammatory condition of the intestines, with its incidence showing a significant year-on-year increase in China. Self-management is becoming increasingly important in the treatment and follow-up of IBD. Numerous studies from Europe and North America have demonstrated that telemedicine can effectively manage disease activity, monitor symptoms, provide education, and improve prognosis. However, its application in China is limited, and there is a lack of high-quality clinical research. This study aims to explore the following objectives:

1. Investigate the level of disease awareness among Chinese IBD patients and their needs related to telemedicine;
2. Develop and preliminarily establish a telemedicine management system and operational process for IBD patients based on a mobile application platform;
3. Clarify the impact of telemedicine on disease activity, quality of life, and healthcare resource utilization among Chinese IBD patients.

DETAILED DESCRIPTION:
To investigate the level of awareness among Chinese IBD (Inflammatory Bowel Disease) patients about their condition and their needs regarding telemedicine, a survey questionnaire has been designed. The questionnaire includes sections on basic knowledge of IBD, treatment methods, daily management, and telemedicine needs. The content of the questionnaire will be discussed and finalized by a team of experts, and then distributed through the Wenjuanxing platform via the WeChat app across multiple centers nationwide, with an expected participation of over 1,000 patients. Additionally, researchers will conduct semi-structured interviews with 50 IBD patients from Changhai Hospital to understand their most concerning symptoms and issues. The results of these interviews will be used to create educational materials for patients.

To construct and operate a telemedicine management system for IBD patients based on the WeChat platform, the following steps will be taken:

1. Establishing Electronic Health Records (EHRs): Each enrolled patient will have an EHR containing personal information, disease history, disease behavior, and treatment details.
2. Health Management Monitoring: Researchers will provide personalized medication and follow-up reminders based on the EHRs. Patients will be encouraged to monitor their health at home, regularly record clinical symptoms, medication, diet, and exercise, and upload this information to the WeChat platform. Self-assessment questionnaires will be distributed periodically via Wenjuanxing to evaluate disease activity, quality of life, sleep, and psychological status, with results recorded in the EHRs.
3. Personalized Recommendations and Interventions: Researchers will assess potential disease risks based on clinical symptoms, self-assessment questionnaires, and medical test results, sending alerts and providing targeted information and interventions.
4. Health Education and Communication: Using results from semi-structured interviews, a health education resource library will be developed, including IBD knowledge, treatment, and daily management in various formats. Weekly personalized education sessions will be provided, and doctor-patient WeChat groups will be established for ongoing interaction, health consultations, and patient discussions.

This section outlines a 12-month, multicenter, randomized controlled clinical trial involving 500 IBD patients across five centers in China. The study aims to explore the impact of WeChat-based telemedicine on disease activity, quality of life, and healthcare resource utilization among IBD patients. Eligible patients will be randomly assigned to either an intervention group or a control group. The intervention group will receive telemedicine management via WeChat, including the establishment of electronic health records, health monitoring, risk alerts, and education, while the control group will receive standard traditional care without additional guidance. All participants will undergo research visits at baseline, 6 months, and 12 months, with colonoscopies required at baseline and 12 months for endoscopic evaluation. Monthly follow-ups via Wenjuanxing will assess healthcare resource utilization. Disease activity (primary endpoint), quality of life, and healthcare resource utilization (secondary endpoints) will be evaluated at baseline, 6 months, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will be diagnosed with IBD based on the diagnostic criteria outlined in the "Consensus on Diagnosis and Treatment of Inflammatory Bowel Disease (2018, Beijing)". The diagnosis will be established by combining clinical symptoms, endoscopic examination results, imaging findings, and histological examination results.
2. Participants must be between the ages of 18 and 75 and provide signed informed consent for the project.
3. Within the two years prior to enrollment, medical records must show at least one instance assessed as an inflammatory active phase (Mayo score ≥ 3 or CDAI score ≥ 150).

Exclusion Criteria:

1. Participants deemed unable to adhere to the study protocol as determined by the investigators.
2. Individuals with a history of surgical treatment for IBD or those scheduled to undergo surgery.
3. Uncontrolled internal medicine or psychiatric disorders.
4. Pregnant individuals or those planning to become pregnant during the enrollment and follow-up period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Disease activity | Six months after enrollment，1 year after enrollment
  Changes in disease activity scores at six months and one year of follow-up after enrollment were assessed. For UC patients, the modified Mayo score (total score 0-12, with higher scores indicating more severe intestinal lesions) was used. For CD patients, the SES-CD score (total score 0-60, with higher scores indicating more severe intestinal lesions) was utilized.

SECONDARY OUTCOMES:
Quality of life assessment | Six months after enrollment，1 year after enrollment
  A multidimensional assessment will be conducted using the widely validated and extensively used patient self-assessment scale, the Simple Quality of Life Questionnaire (IBDQ). This scale consists of 32 selected health-related questions (total score 32-224, with higher scores indicating better quality of life).
Psychological assessment | Six months after enrollment，1 year after enrollment
  The assessment is conducted using the Hospital Anxiety and Depression Scale (HADS), which consists of 14 emotional questions. The total score ranges from 0 to 42, with higher scores indicating more severe psychological distress in patients.
Utilization rate of medical resources | Each month within the 1 year of enrollment
  The assessment of healthcare resource utilization will be conducted through a self-administered questionnaire. Follow-up questionnaires will be administered via the WeChat Questionnaire Star platform in the 1st, 2nd, 3rd, 4th, 5th, 7th, 8th, 9th, 10th, and 11th months to evaluate healthcare resource utilization patterns. This questionnaire has been developed through an extensive review of the literature and discussions with relevant experts. Its key components include total number of medical visits, IBD-related hospitalizations, emergency room visits, outpatient visits, endoscopic examinations, and telemedicine consultations.（The more frequently the relevant information is filled out, the lower the utilization of medical resources.）
Ratio of reduced IBD flare-up episodes | 1 year after enrollment
  The proportion of patients with reduced IBD flare-ups (one year before and after enrollment). IBD patients in a flare-up phase within one month after enrollment were excluded.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, Professor, Study Director — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seyed Tabib NS, Madgwick M, Sudhakar P, Verstockt B, Korcsmaros T, Vermeire S. Big data in IBD: big progress for clinical practice. Gut. 2020 Aug;69(8):1520-1532. doi: 10.1136/gutjnl-2019-320065. Epub 2020 Feb 28. PMID 32111636
- [Background] Mak WY, Zhao M, Ng SC, Burisch J. The epidemiology of inflammatory bowel disease: East meets west. J Gastroenterol Hepatol. 2020 Mar;35(3):380-389. doi: 10.1111/jgh.14872. Epub 2019 Nov 24. PMID 31596960
- [Background] Burisch J, Zhao M, Odes S, De Cruz P, Vermeire S, Bernstein CN, Kaplan GG, Duricova D, Greenberg D, Melberg HO, Watanabe M, Ahn HS, Targownik L, Pittet VEH, Annese V, Park KT, Katsanos KH, Hoivik ML, Krznaric Z, Chaparro M, Loftus EV Jr, Lakatos PL, Gisbert JP, Bemelman W, Moum B, Gearry RB, Kappelman MD, Hart A, Pierik MJ, Andrews JM, Ng SC, D'Inca R, Munkholm P. The cost of inflammatory bowel disease in high-income settings: a Lancet Gastroenterology & Hepatology Commission. Lancet Gastroenterol Hepatol. 2023 May;8(5):458-492. doi: 10.1016/S2468-1253(23)00003-1. Epub 2023 Mar 2. PMID 36871566
- [Background] Hulme JB, Bain B, Hardin M, McKinnon A, Waldron D. The influence of adaptive seating devices on vocalization. J Commun Disord. 1989 Apr;22(2):137-45. doi: 10.1016/0021-9924(89)90030-0. PMID 2723144
- [Background] Singh A, Koenen B, Kirby DF. Bariatric Surgery and Its Complications in Inflammatory Bowel Disease Patients. Inflamm Bowel Dis. 2020 Jul 17;26(8):1155-1165. doi: 10.1093/ibd/izz246. PMID 31626698
- [Background] Gold SL, Rabinowitz LG, Manning L, Keefer L, Rivera-Carrero W, Stanley S, Sherman A, Castillo A, Tse S, Hyne A, Matos K, Cohen B, Grinspan A, Colombel JF, Sands BE, Dubinsky MC, Ungaro RC. High Prevalence of Malnutrition and Micronutrient Deficiencies in Patients With Inflammatory Bowel Disease Early in Disease Course. Inflamm Bowel Dis. 2023 Mar 1;29(3):423-429. doi: 10.1093/ibd/izac102. PMID 35590456
- [Background] Bai Y, Peng J, Gao J, Zou DW, Li ZS. Epidemiology of lower gastrointestinal bleeding in China: single-center series and systematic analysis of Chinese literature with 53,951 patients. J Gastroenterol Hepatol. 2011 Apr;26(4):678-82. doi: 10.1111/j.1440-1746.2010.06586.x. PMID 21083610
- [Background] Turner D, Ricciuto A, Lewis A, D'Amico F, Dhaliwal J, Griffiths AM, Bettenworth D, Sandborn WJ, Sands BE, Reinisch W, Scholmerich J, Bemelman W, Danese S, Mary JY, Rubin D, Colombel JF, Peyrin-Biroulet L, Dotan I, Abreu MT, Dignass A; International Organization for the Study of IBD. STRIDE-II: An Update on the Selecting Therapeutic Targets in Inflammatory Bowel Disease (STRIDE) Initiative of the International Organization for the Study of IBD (IOIBD): Determining Therapeutic Goals for Treat-to-Target strategies in IBD. Gastroenterology. 2021 Apr;160(5):1570-1583. doi: 10.1053/j.gastro.2020.12.031. Epub 2021 Feb 19. PMID 33359090
- [Background] Colombel JF, Narula N, Peyrin-Biroulet L. Management Strategies to Improve Outcomes of Patients With Inflammatory Bowel Diseases. Gastroenterology. 2017 Feb;152(2):351-361.e5. doi: 10.1053/j.gastro.2016.09.046. Epub 2016 Oct 5. PMID 27720840
- [Background] Yu Q, Zhu C, Feng S, Xu L, Hu S, Chen H, Chen H, Yao S, Wang X, Chen Y. Economic Burden and Health Care Access for Patients With Inflammatory Bowel Diseases in China: Web-Based Survey Study. J Med Internet Res. 2021 Jan 5;23(1):e20629. doi: 10.2196/20629. PMID 33399540
- [Background] Szigethy EM, Allen JI, Reiss M, Cohen W, Perera LP, Brillstein L, Cross RK, Schwartz DA, Kosinski LR, Colton JB, LaRusso E, Atreja A, Regueiro MD. White Paper AGA: The Impact of Mental and Psychosocial Factors on the Care of Patients With Inflammatory Bowel Disease. Clin Gastroenterol Hepatol. 2017 Jul;15(7):986-997. doi: 10.1016/j.cgh.2017.02.037. Epub 2017 Mar 12. PMID 28300693
- [Background] Colombel JF, Panaccione R, Bossuyt P, Lukas M, Baert F, Vanasek T, Danalioglu A, Novacek G, Armuzzi A, Hebuterne X, Travis S, Danese S, Reinisch W, Sandborn WJ, Rutgeerts P, Hommes D, Schreiber S, Neimark E, Huang B, Zhou Q, Mendez P, Petersson J, Wallace K, Robinson AM, Thakkar RB, D'Haens G. Effect of tight control management on Crohn's disease (CALM): a multicentre, randomised, controlled phase 3 trial. Lancet. 2017 Dec 23;390(10114):2779-2789. doi: 10.1016/S0140-6736(17)32641-7. Epub 2017 Oct 31. PMID 29096949
- [Background] Kane SV, Cohen RD, Aikens JE, Hanauer SB. Prevalence of nonadherence with maintenance mesalamine in quiescent ulcerative colitis. Am J Gastroenterol. 2001 Oct;96(10):2929-33. doi: 10.1111/j.1572-0241.2001.04683.x. PMID 11693328
- [Background] Levine A, Rhodes JM, Lindsay JO, Abreu MT, Kamm MA, Gibson PR, Gasche C, Silverberg MS, Mahadevan U, Boneh RS, Wine E, Damas OM, Syme G, Trakman GL, Yao CK, Stockhamer S, Hammami MB, Garces LC, Rogler G, Koutroubakis IE, Ananthakrishnan AN, McKeever L, Lewis JD. Dietary Guidance From the International Organization for the Study of Inflammatory Bowel Diseases. Clin Gastroenterol Hepatol. 2020 May;18(6):1381-1392. doi: 10.1016/j.cgh.2020.01.046. Epub 2020 Feb 15. PMID 32068150
- [Background] Mikocka-Walus A, Knowles SR, Keefer L, Graff L. Controversies Revisited: A Systematic Review of the Comorbidity of Depression and Anxiety with Inflammatory Bowel Diseases. Inflamm Bowel Dis. 2016 Mar;22(3):752-62. doi: 10.1097/MIB.0000000000000620. PMID 26841224
- [Background] Ahmed W, Taft TH, Charabaty A. Social media in inflammatory bowel disease: the patient and physician perspective. Curr Opin Gastroenterol. 2021 Jul 1;37(4):328-335. doi: 10.1097/MOG.0000000000000742. PMID 33859103
- [Background] Reich J, Guo L, Groshek J, Weinberg J, Chen W, Martin C, Long MD, Farraye FA. Social Media Use and Preferences in Patients With Inflammatory Bowel Disease. Inflamm Bowel Dis. 2019 Feb 21;25(3):587-591. doi: 10.1093/ibd/izy280. PMID 30203036
- [Background] Song S, Zhang Y, Yu B. Interventions to support consumer evaluation of online health information credibility: A scoping review. Int J Med Inform. 2021 Jan;145:104321. doi: 10.1016/j.ijmedinf.2020.104321. Epub 2020 Nov 1. PMID 33202372
- [Background] Sun Y, Zhang Y, Gwizdka J, Trace CB. Consumer Evaluation of the Quality of Online Health Information: Systematic Literature Review of Relevant Criteria and Indicators. J Med Internet Res. 2019 May 2;21(5):e12522. doi: 10.2196/12522. PMID 31045507
- [Background] van der Marel S, Duijvestein M, Hardwick JC, van den Brink GR, Veenendaal R, Hommes DW, Fidder HH. Quality of web-based information on inflammatory bowel diseases. Inflamm Bowel Dis. 2009 Dec;15(12):1891-6. doi: 10.1002/ibd.20976. Epub 2009 May 21. PMID 19462423
- [Background] Sato H. [On the manual dexterity and behavior of daily living of children]. Ann Physiol Anthropol. 1987 Jul;6(3):171-4. No abstract available. Japanese. PMID 3675775
- [Background] Scanfeld D, Scanfeld V, Larson EL. Dissemination of health information through social networks: twitter and antibiotics. Am J Infect Control. 2010 Apr;38(3):182-8. doi: 10.1016/j.ajic.2009.11.004. PMID 20347636
- [Background] Ross JR. Veneered osseous graft. Case report and technique. J Tenn Dent Assoc. 1990 Jul;70(3):14-6. PMID 2214749
- [Background] Mason AN. The Most Important Telemedicine Patient Satisfaction Dimension: Patient-Centered Care. Telemed J E Health. 2022 Aug;28(8):1206-1214. doi: 10.1089/tmj.2021.0322. Epub 2021 Dec 8. PMID 34882032
- [Background] Pengput A, Schwartz DG. Telemedicine in Southeast Asia: A Systematic Review. Telemed J E Health. 2022 Dec;28(12):1711-1733. doi: 10.1089/tmj.2021.0516. Epub 2022 Apr 12. PMID 35417250
- [Background] Erdur H, Weber JE, Angermaier A, Kinze S, Sotoodeh A, Gorski C, Bollweg K, Ernst S, Kandil FI, Behrens J, Ganeshan R, Keysers A, Kotlarz-Bottcher M, Peters D, Schlemm L, Stangenberg-Gliss K, Witt C, Hennig B, Reber KC, Schneider U, Franke C, Schmehl I, Straub HB, Floel A, Theen S, Endres M, Kurth T, Audebert HJ. A Managed Care System with Telemedicine Support for Neurological Emergencies. Ann Neurol. 2023 Mar;93(3):511-521. doi: 10.1002/ana.26556. Epub 2022 Dec 2. PMID 36401341
- [Background] Tilden DR, Datye KA, Moore DJ, French B, Jaser SS. The Rapid Transition to Telemedicine and Its Effect on Access to Care for Patients With Type 1 Diabetes During the COVID-19 Pandemic. Diabetes Care. 2021 Jun;44(6):1447-1450. doi: 10.2337/dc20-2712. Epub 2021 Apr 13. PMID 33849938
- [Background] Chow CK, Redfern J, Hillis GS, Thakkar J, Santo K, Hackett ML, Jan S, Graves N, de Keizer L, Barry T, Bompoint S, Stepien S, Whittaker R, Rodgers A, Thiagalingam A. Effect of Lifestyle-Focused Text Messaging on Risk Factor Modification in Patients With Coronary Heart Disease: A Randomized Clinical Trial. JAMA. 2015 Sep 22-29;314(12):1255-63. doi: 10.1001/jama.2015.10945. PMID 26393848
- [Background] de Jong MJ, van der Meulen-de Jong AE, Romberg-Camps MJ, Becx MC, Maljaars JP, Cilissen M, van Bodegraven AA, Mahmmod N, Markus T, Hameeteman WM, Dijkstra G, Masclee AA, Boonen A, Winkens B, van Tubergen A, Jonkers DM, Pierik MJ. Telemedicine for management of inflammatory bowel disease (myIBDcoach): a pragmatic, multicentre, randomised controlled trial. Lancet. 2017 Sep 2;390(10098):959-968. doi: 10.1016/S0140-6736(17)31327-2. Epub 2017 Jul 14. PMID 28716313
- [Background] George LA, Dominic MR, Cross RK. Integration of telemedicine into clinical practice for inflammatory bowel disease. Curr Opin Gastroenterol. 2020 Jul;36(4):304-309. doi: 10.1097/MOG.0000000000000647. PMID 32398568
- [Background] Reigada LC, Satpute A, Hoogendoorn CJ, Cohen BH, Lai J, Bao R, Dubinsky MC, Benkov KJ. Patient-reported Anxiety: A Possible Predictor of Pediatric Inflammatory Bowel Disease Health Care Use. Inflamm Bowel Dis. 2016 Sep;22(9):2127-33. doi: 10.1097/MIB.0000000000000864. PMID 27482980
- [Background] Elkjaer M, Shuhaibar M, Burisch J, Bailey Y, Scherfig H, Laugesen B, Avnstrom S, Langholz E, O'Morain C, Lynge E, Munkholm P. E-health empowers patients with ulcerative colitis: a randomised controlled trial of the web-guided 'Constant-care' approach. Gut. 2010 Dec;59(12):1652-61. doi: 10.1136/gut.2010.220160. PMID 21071584
- [Background] Cross RK, Cheevers N, Rustgi A, Langenberg P, Finkelstein J. Randomized, controlled trial of home telemanagement in patients with ulcerative colitis (UC HAT). Inflamm Bowel Dis. 2012 Jun;18(6):1018-25. doi: 10.1002/ibd.21795. Epub 2011 Jun 17. PMID 21688350
- [Background] Harvey RF, Bradshaw JM. A simple index of Crohn's-disease activity. Lancet. 1980 Mar 8;1(8167):514. doi: 10.1016/s0140-6736(80)92767-1. No abstract available. PMID 6102236
- [Background] Walmsley RS, Ayres RC, Pounder RE, Allan RN. A simple clinical colitis activity index. Gut. 1998 Jul;43(1):29-32. doi: 10.1136/gut.43.1.29. PMID 9771402
- [Background] Cross RK, Langenberg P, Regueiro M, Schwartz DA, Tracy JK, Collins JF, Katz J, Ghazi L, Patil SA, Quezada SM, Beaulieu D, Horst SN, Russman K, Riaz M, Jambaulikar G, Sivasailam B, Quinn CC. A Randomized Controlled Trial of TELEmedicine for Patients with Inflammatory Bowel Disease (TELE-IBD). Am J Gastroenterol. 2019 Mar;114(3):472-482. doi: 10.1038/s41395-018-0272-8. PMID 30410041